CLINICAL TRIAL: NCT02049619
Title: Do Pharyngeal Packs During Orthognathic Surgery Reduce Postoperative Nausea and Vomiting. A Prospective Randomized Double Blind Clinical Trial.
Brief Title: Do Pharyngeal Packs During Orthognathic Surgery Reduce Postoperative Nausea and Vomiting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Xia Zhang, assistant professor, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UMC-PONV
Record Dates: First submitted 2014-01-27; First posted 2014-01-30 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Nausea; Vomiting
Keywords: Pharyngeal pack; Nausea; Vomiting; orthognathic surgery; maxillary osteotomy
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Following endotracheal intubation, no pharyngeal pack was inserted into the hypopharynx.
- pharyngeal pack (Experimental): Following endotracheal intubation, one saline soaked, gauze pharyngeal pack was inserted into the hypopharynx under direct vision using McGill's forceps. The packs were tied to the endotracheal tube and their placements were documented on the scrub nurse's count board.
  Interventions: Device: pharyngeal pack

INTERVENTIONS:
Device: pharyngeal pack — Following endotracheal intubation, one saline soaked, gauze pharyngeal pack was inserted into the hypopharynx under direct vision using McGill's forceps. The packs were tied to the endotracheal tube and their placements were documented on the scrub nurse's count board.
  Arms: pharyngeal pack

SUMMARY:
The purpose of this study is to determine whether pharyngeal packs can reduce nausea and vomiting in patients undergoing orthognathic surgery.

DETAILED DESCRIPTION:
Post-operative nausea and vomiting (PONV) is one of the most frequent and distressing complications of anesthesia. Patients often rate that PONV is worse than postoperative pain. PONV alone is one of the leading causes for delayed discharge and unpleasant experiments. Although PONV is not always life-threatening, persistent cases can result in dehydration, esophageal rupture, aspiration and potential death. The massive ingested blood and the additional issue of an altered diet (full liquids) due to a short period of jaw immobilization may be associated with a higher prevalence of PONV after orthognathic surgeries.

Although most of antiemetic drugs can help prevent PONV, they cannot preclude vomiting resulting from irritating gastrointestinal stimuli such as blood in the stomach. Pharyngeal packs are thought to prevent the ingestion and aspiration of blood, cartilage and bone fragments during oral and maxillofacial surgeries. Whether pharyngeal packs can reduce the incidence of PONV is controversial. It is reported that pharyngeal packs are recommended for the purpose of preventing PONV in nasal surgeries. However, some authors suggest that pharyngeal packs have no impact on PONV or the prevalence of PONV is doubled during routine nasal surgeries. However, the population size in these studies is relatively small and the trials have significant methodological weakness. None of these trials totally addressed the issue of the pharyngeal packs on the PONV following nasal surgeries. Moreover, these studies include different types of nasal surgeries, not all of which can be assumed to have equivalent bleeding potential.

Orthognathic surgeries performed maxillary and mandibular osteotomies and are assumed to involve massive blood loss. Orofacial swelling and swallowing blood is common in the early postoperative period after orthognathic surgeries. Whether pharyngeal packs can reduce the swallowing blood and PONV is unknown. Thus, The objective of this study is to determine whether pharyngeal packs can reduce nausea and vomiting in patients undergoing orthognathic surgery.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective orthognathic surgery
* age 18-50 year olds
* signed informed consent

Exclusion Criteria:

* pregnant women
* past history of oesophageal surgery, oesophageal varices or stricture,
* patients who have received antiemetic medication in the 24 hours before surgery
* emergency surgery
* prior history of motion sickness and/or PONV, vertigo or migraine headaches

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
the incidence and severity of any nausea, emetic episodes (retching or vomiting), or both (i.e., postoperative nausea and vomiting) during the first 24 postoperative hours. | the first 24 postoperative hours
  The primary outcome measure was the incidence and severity of any nausea, emetic episodes (retching or vomiting), or both (i.e., postoperative nausea and vomiting) during the first 24 postoperative hours. After the 2nd, 4th, 6th and 24th postoperative hours, trained investigators who were fully blinded to the intraoperative management and random treatment assignments recorded the number of emetic episodes, the volume of vomiting, and the time each one occurred. 0 represented no PONV and 10 represented the most severe PONV possible.

SECONDARY OUTCOMES:
The incidence and severity of throat pain | the first 24 postoperative hours
  0 represented no throat pain and 10 represented the most severe throat pain possible.
the incidence of oral mucosal injury | the first 24 postoperative hours
satisfactory scores of patients | the first 24 postoperative hours
  0 represented that patients are not satisfactory with the anesthesia and 10 represented that patients are very satisfactory with the anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: xia zhang, MD, Principal Investigator — School & Hospital of Stomatology, China Medical University, China
Locations (1):
- School & Hospital of Stomatology, China Medical University, Shenyang, Liaoning, China